CLINICAL TRIAL: NCT06397820
Title: Relation Between Artificial Intelligence (AI)-Assisted Quantitative Coronary Angiography and Positron Emission Tomography-Derived Myocardial Blood Flow
Brief Title: Relation Between AI-QCA and Cardiac PET
Acronym: AI-CARPET
Status: Completed | Type: Observational
Sponsor: Chonnam National University Hospital (Other)
Responsible Party: Principal Investigator, Seung Hun Lee, Assistant Professor, Chonnam National University Hospital
Other Study IDs: CNUH-AI-CARPET
Record Dates: First submitted 2024-04-30; First posted 2024-05-03 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Coronary Artery Disease; Coronary Artery Stenosis
Keywords: Invasive coronary angiography; Cardaic positron Emission Tomography; Artificial Intelligence; Quantitative Coronary Angiography
MeSH Terms: conditions — Coronary Artery Disease; Coronary Stenosis | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Positive for PET-derived indexes: Patients who had decreased stress myocardial blood flow (MBF) or relative flow ratio (RFR) on PET
  Interventions: Device: Percutaneous coronary intervention (PCI)
- Negative for PET-derived indexes: Patients who had preserved stress myocardial blood flow (MBF) or relative flow ratio (RFR) on PET

INTERVENTIONS:
Device: Percutaneous coronary intervention (PCI) — Revascularization by percutaneous coronary intervention for vessels with decreased PET-derived flow indexes
  Groups: Positive for PET-derived indexes

SUMMARY:
The aim of the study is to evaluate the clinical implications of artificial Intelligence (AI)-assisted quantitative coronary angiography (QCA) and positron emission tomography (PET)-derived myocardial blood flow in clinically indicated patients.

DETAILED DESCRIPTION:
Percutaneous coronary angiography (CAG) is a standard method for evaluating coronary artery disease. Traditionally, a reduction in the luminal diameter of the coronary arteries by 50% or more during angiography has been considered a significant stenotic lesion. However, the assessment of coronary artery stenosis is usually based on visual estimation by the operator in daily routine clinical practice, which interferes with the objective evaluation.

Quantitative coronary angiography (QCA) has been developed to overcome this limitation. This technique involves the software-based analysis of coronary images obtained through CAG. The previous study showed that there was low concordance between the QCA and visual estimation of coronary artery stenosis (Kappa=0.63) and a reclassification rate of approximately 20%. Furthermore, visual assessments tended to overestimate the degree of coronary artery stenosis, particularly in complex lesions such as bifurcation lesions.

However, there are some limitations to adopting QCA in our daily routine practice. The QCA cannot analyze coronary images on-site and is not fully automated, requiring manual adjustments by humans. Recent advancements have led to the development of artificial intelligence (AI)-based QCA software, which achieves complete automation in the analysis process and provides real-time objective evaluations of coronary artery stenosis.

This study aims to examine the clinical significance of AI-QCA by assessing the correlation between the degree of coronary stenosis detected by AI-QCA and myocardial blood flow abnormalities observed in 13NH3-Ammonia PET scans in patients with coronary artery disease.

ELIGIBILITY:
Inclusion criteria

1. Subject must be ≥18 years
2. Patients suspected with CAD or ischemic heart disease
3. Patients undergoing CAG and cardiac PET for evaluation of severity of coronary artery disease

Exclusion criteria

1. Poor imaging quality of CAG and PET which were not available for core-lab analysis
2. Chronic total occlusion
3. Time interval was more than >3 months between CAG and PET
4. History of coronary artery bypass grafting
5. History of acute myocardial infarction or recent myocardial infarction
6. Heart failure (left ventricular ejection fraction <40%)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with suspected coronary artery disease (CAD) undergoing invasive coronary angiography (CAG) and clinically indicated for cardiac PET assessment.
Sampling Method: Probability Sample
Enrollment: 168 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Correlation between diameter stenosis by AI-QCA and PET-driven RFR | Immediate after AI-QCA and PET exams
  Performance of AI-QCA predicting for PET-driven RFR
Correlation between diameter stenosis by AI-QCA and PET-driven stress MBF | Immediate after AI-QCA and PET exams
  Performance of AI-QCA predicting for PET-driven stress MBF

SECONDARY OUTCOMES:
Correlation between diameter stenosis by AI-QCA and PET-driven coronary flow reserve (CFR) | Immediate after AI-QCA and PET exams
  Performance of AI-QCA predicting for PET-driven CFR
Correlation between diameter stenosis by AI-QCA and PET-driven coronary flow capacity (CFC) | Immediate after AI-QCA and PET exams
  Performance of AI-QCA predicting for PET-driven CFC
Correlation between diameter stenosis by AI-QCA and PET-driven semi-quantitative markers of ischemia | Immediate after AI-QCA and PET exams
  Performance of AI-QCA predicting for PET-driven semi-quantitative markers of ischemia
All-cause death | 1 year after last patient enrollment
  All-cause death
Cardiovascular death | 1 year after last patient enrollment
  Cardiovascular death
Myocardial infarction | 1 year after last patient enrollment
  Any myocardial infarction, defined by Forth Universal definition of myocardial infarction
Rate of target lesion revascularization | 1 year after last patient enrollment
  Target lesion revascularization
Rate of target vessel revascularization | 1 year after last patient enrollment
  Target vessel revascularization
Rate of any revascularization | 1 year after last patient enrollment
  Any revascularization
Rate of stent thrombosis | 1 year after last patient enrollment
  Definite or probable stent thrombosis, defined by ARC II definition
Rate of cerebrovascular accident | 1 year after last patient enrollment
  Cerebrovascular accident
Major adverse cerebrocardiovascular event (MACCE) | 1 year after last patient enrollment
  A composite of death, myocardial infarction, any revascularization, and cerebrovascular accident

CONTACTS AND LOCATIONS:
Overall Officials: Sang-Geon Cho, MD, PhD, Principal Investigator — Chonnam National University Hospital; Seung Hun Lee, MD, PhD, Principal Investigator — Chonnam National University Hospital
Locations (1):
- Chonnam National University Hospital, Gwangju, South Korea

IPD SHARING:
Plan to Share IPD: Yes
After publication of main paper, de-identified data will be shared upon reasonable requests after discussion by Executive Committee.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After publication of main paper.
Access Criteria: Executive Committee will discuss to share the de-identified data upon reasonable requests.